CLINICAL TRIAL: NCT03321175
Title: Evaluation the Impact of Subcutaneous Irrigation on Wound Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berna Aslan Cetin, Attending physician,ObGyn, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2017/219
Record Dates: First submitted 2017-10-22; First posted 2017-10-25 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Cesarean Section; Complications, Wound, Hematoma
Keywords: Wound; infection; cesarean section
MeSH Terms: conditions — Wounds and Injuries; Hematoma; Infections

STUDY DESIGN:
Intervention Model Description: Randomization will be performed by an online software. Randomized cards will be in sealed envelopes and will be open by surgeon at the time of surgery.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subcutaneous irrigaton (Experimental): Patients will receive 200 cc subcutaneous saline irrigation before skin incision closure.
  Interventions: Other: subcutaneous saline irrigation
- Subcutaneous no irrigation (No Intervention): Patients will not receive subcutaneous saline irrigation before skin incision closure.

INTERVENTIONS:
Other: subcutaneous saline irrigation — 200 cc saline irrigation
  Arms: Subcutaneous irrigaton

SUMMARY:
to evaluate the effect of subcutaneous irrigation on wound complications

DETAILED DESCRIPTION:
Cesarean section is the most common abdominal operation performed worldwide. As with every other surgical procedure, it is sometimes accompanied by surgical complications. Wound complications are encountered in approximately 5% of women that undergo CS and include haematomas, seromas and infection. To evaluate the effects and benefits of subcutaneous irrigation during cesarean section we decide to conduct this randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40, undergoing cesarean section

Exclusion Criteria:

* patients with systemical disease, body mass index>30

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients undergoing cesarean section
Enrollment: 185 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
wound complications | 1 week
  wound complications will be evaluated 1 week after the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni SSTRH, Istanbul, Turkey (Türkiye)